CLINICAL TRIAL: NCT05081726
Title: Functional MRI in Older People Following Hip Fracture Surgery: a Feasibility Study
Brief Title: fMRI Feasibility Older Hip Fracture Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 19087
Record Dates: First submitted 2020-02-28; First posted 2021-10-18 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Magnetic Resonance Imaging; Hip Fractures; Postoperative Delirium
Keywords: older people; postoperative delirium; Functional MRI
MeSH Terms: conditions — Hip Fractures; Emergence Delirium | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Never had delirium: Older people recovering from hip fracture surgery who did not have postoperative delirium
  Interventions: Diagnostic Test: Functional MRI
- Recovered delirium: Older people recovering from hip fracture surgery who experienced delirium which has resolved
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — Series of MRI scans of the brain

SUMMARY:
An assessment of the feasibility of structural and functional magnetic resonance imaging (MRI) brain scans in older people who have recovered from and older people who never had delirium after hip fracture surgery

DETAILED DESCRIPTION:
Postoperative delirium, an acute sate of confusion occurs with higher frequency in older people. Hip fracture surgery is a procedure associated with an increased risk of postoperative delirium.

In the study the feasibility of achieving structure and functional connectivity imaging of the brain, using magnetic resonance imaging, in older people who are recovering from hip fracture surgery will be assessed.

People who have recovered from post operative delirium and people who did not have postoperative delirium will be included.

ELIGIBILITY:
Inclusion Criteria:Age

* Age ≥ 65 years
* Cognitively intact
* primary admission for hip fracture surgery

Exclusion Criteria:

* Cognitive impairment
* Less than moderate level of activities of daily living
* History of neurosurgery/significant head trauma
* Acutely unwell/moribund
* Presence of neurological diseases including overt stroke, dementia, multiple sclerosis, Parkinson's disease, intracranial tumours and other significant neurologic disorders.
* Postural or movement disorders likely to impede MRI scan
* Contraindications to MRI
* Complex fractures/multiple injuries

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older people recovering from hip fracture surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-07-04 (Estimated); Primary Completion 2022-09-02 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MRI in older people following hip fracture surgery assessed by tolerability of transfer to scanner and the scanning process | From time of consent to day after MRI scan which is up to 5 days
  The feasibility of transferring participants to and achieving structural and functional MRI scans. Specifically we will assess the number of participants in whom scans were successfully achieved

SECONDARY OUTCOMES:
Abnormalities of functional connectivity | Up to one month after scans have been achieved
  Identify any differences in functional connectivity between the resolved delirium and the never delirium MRI scans
Pain assessment. | From immediately prior to transfer to the MRI suite until return to own hospital bed which is approximately 2 hours
  An assessment of baseline pain levels and then repeat assessments of pain during transfer and the MRI scanning process using the numerical pain rating scale
Actual times taken to achieve scans | Up to 60 minutes
  An assessment of unforeseen constraints on time taken to scan
Participant feedback | Two occassions. The first immediately after return from the MRI scan suite. The second will occur the day after scanning. Each will take 5 minutes.
  The participant experience will be explored via verbal feedback which will be documented by the accompanying researcher

CONTACTS AND LOCATIONS:
Overall Officials: Rob Dineen, PhD, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
Incidental findings in participants who give consent for sharing of these with their physician, will be communicated to the general practitioner for further action if required.